CLINICAL TRIAL: NCT03330275
Title: Evaluating the Impact of JJVC Senofilcon A - Based Contact Lens With New UV-blocker on Day and Night Driving Performance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5830
Record Dates: First submitted 2017-10-17; First posted 2017-11-06 (Actual); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Visual Performance
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Test/Control 1/Control 2 (Experimental): Subjects will be randomized to 1 of 3 lenses (Test/Control 1/Control 2). Subjects will also be randomized to (1) Sequence of driving time (Day and Night) and (2) Driving Route (A, B, C). Hazard and pedestrian locations will be randomized for each driving route.
  Interventions: Device: Investigational Contact Lens; Device: Commercial ACUVUE OASYS; Device: Commercial ACUVUE OASYS and Spectacles
- Test/Control 2/Control 1 (Experimental): Subjects will be randomized to 1 of 3 lenses (Test/Control 2/Control 1). Subjects will also be randomized to (1) Sequence of driving time (Day and Night) and (2) Driving Route (A, B, C). Hazard and pedestrian locations will be randomized for each driving route.
  Interventions: Device: Investigational Contact Lens; Device: Commercial ACUVUE OASYS; Device: Commercial ACUVUE OASYS and Spectacles
- Control 1/Test/Control 2 (Experimental): Subjects will be randomized to 1 of 3 lenses (Control 1/Test/Control 2). Subjects will also be randomized to (1) Sequence of driving time (Day and Night) and (2) Driving Route (A, B, C). Hazard and pedestrian locations will be randomized for each driving route.
  Interventions: Device: Investigational Contact Lens; Device: Commercial ACUVUE OASYS; Device: Commercial ACUVUE OASYS and Spectacles
- Control 1/Control 2/Test (Experimental): Subjects will be randomized to 1 of 3 lenses (Control 1/Control 2/Test). Subjects will also be randomized to (1) Sequence of driving time (Day and Night) and (2) Driving Route (A, B, C). Hazard and pedestrian locations will be randomized for each driving route.
  Interventions: Device: Investigational Contact Lens; Device: Commercial ACUVUE OASYS; Device: Commercial ACUVUE OASYS and Spectacles
- Control 2/Test/Control 1 (Experimental): Subjects will be randomized to 1 of 3 lenses (Control 2/Test/Control 1). Subjects will also be randomized to (1) Sequence of driving time (Day and Night) and (2) Driving Route (A, B, C). Hazard and pedestrian locations will be randomized for each driving route.
  Interventions: Device: Investigational Contact Lens; Device: Commercial ACUVUE OASYS; Device: Commercial ACUVUE OASYS and Spectacles
- Control 2/Control 1/Test (Experimental): Subjects will be randomized to 1 of 3 lenses (Control 2/Control 1/Test). Subjects will also be randomized to (1) Sequence of driving time (Day and Night) and (2) Driving Route (A, B, C). Hazard and pedestrian locations will be randomized for each driving route.
  Interventions: Device: Investigational Contact Lens; Device: Commercial ACUVUE OASYS; Device: Commercial ACUVUE OASYS and Spectacles

INTERVENTIONS:
Device: Investigational Contact Lens — JJVC senofilcon A-based contact lens with new UV-blocker
  Other Names: Test
Device: Commercial ACUVUE OASYS — senofilcon A
  Other Names: Control 1
Device: Commercial ACUVUE OASYS and Spectacles — Senofilcon A and Spectacles
  Other Names: Control 2

SUMMARY:
This is a bilateral, non-dispensing, randomized, subject masked, four visits, 3-period by 3- treatment crossover study. The objective of this study is to evaluate the effect of JJVC senofilcon A - based contact lens with new UV-blocker on vision and driving performance in both daytime and nighttime lighting under real world driving conditions. This will be achieved through field-based driving studies on a closed-road driving circuit at night and during the day. Quantitative methods will be used to assess vision and driving performance under a range of challenging conditions and appropriate masking, order of testing, randomization and control conditions will be used.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 20 and 49 (inclusive) years of age at the time of screening.
  4. Presbyopic subjects must be habitual wearers of distance vision correction in both eyes.
  5. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 through -6.00 D (inclusive) in each eye.
  6. The subject's refractive cylinder must be ≤ 1.00 D in each eye.
  7. Have spherocylindrical best corrected visual acuity of 20/20 or better in each eye.
  8. Be a current soft contact lens wearer in both eyes, defined as at least 5 days per week and 6 hours per day averaged over the past 30 days.
  9. Hold a current Open driver's license
  10. Be a regular driver (at least once per week)
  11. Have at least one year of driving experience

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear, pupil size or accommodation.
  4. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  5. History of binocular vision abnormality or strabismus
  6. Any current use of ocular medication
  7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
  8. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA slit lamp biomicroscopy scale
  9. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear
  10. Employee of clinical site (e.g., Investigator, Coordinator, Technician)

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Queensland University of Technology, School of Optometry and Vision Science, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buch JR, Toubouti Y, Cannon J. Randomized Crossover Trial Evaluating the Impact of Senofilcon A Photochromic Lens on Driving Performance. Optom Vis Sci. 2020 Jan;97(1):15-23. doi: 10.1097/OPX.0000000000001466. PMID 31895273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 subjects were enrolled into this study. All enrolled subjects met all eligibility criteria and were dispensed a study lens. Of the dispensed subjects, all 24 completed the study.
Pre-assignment Details: A 2X2 William's crossover design was utilized for visit 1. A 3X3 William's Crossover design was utilized for visits 2, 3 and 4.
Groups:
- Test/Control1: Subjects that were randomized to receive the Test lens during period 1 of visit 1 and the Control 1 lens during period 2 of visit 1.
- Control1/Test: Subjects that were randomized to receive the Control 1 lens during period 1 of visit 1 and the Test lens during period 2 of visit 1.
- Test/Control2: Subjects that were randomized to receive the Test lens during period 1 of visit 1 and the Control 2 lens during period 2 of visit 1.
- Control2/Test: Subjects that were randomized to receive the Control 2 lens during period 1 of visit 1 and the Test lens during period 2 of visit 1.
- Test/Control1/Control2: Subjects that were randomized to receive the Test lens during period 1, the Control 1 lens during period 2 and the Control 2 lens during period 3. This applies to visits 2, 3 and 4.
- Test/Control2/Control1: Subjects that were randomized to receive the Test lens during period 1, the Control 2 lens during period 2 and the Control 1 lens during period 3. This applies to visits 2, 3 and 4.
- Control1/Control2/Test: Subjects that were randomized to receive the Control 1 lens during period 1, the Control 2 lens during period 2 and the Test lens during period 3. This applies to visits 2, 3 and 4.
- Control1/Test/Control2: Subjects that were randomized to receive the Control 1 lens during period 1, the Test lens during period 2 and the Control 2 lens during period 3. This applies to visits 2, 3 and 4.
- Control2/Control1/Test: Subjects that were randomized to receive the Control 2 lens during period 1, the Control 1 lens during period 2 and the Test lens during period 3. This applies to visits 2, 3 and 4.
- Control2/Test/Control1: Subjects that were randomized to receive the Control 2 lens during period 1, the Test lens during period 2 and the Control 1 lens during period 3. This applies to visits 2, 3 and 4.
Period: Visit 1 - Period 1
Arm/Group | Test/Control1 | Control1/Test | Test/Control2 | Control2/Test | Test/Control1/Control2 | Test/Control2/Control1 | Control1/Control2/Test | Control1/Test/Control2 | Control2/Control1/Test | Control2/Test/Control1
Started | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 1 - Period 2
Arm/Group | Test/Control1 | Control1/Test | Test/Control2 | Control2/Test | Test/Control1/Control2 | Test/Control2/Control1 | Control1/Control2/Test | Control1/Test/Control2 | Control2/Control1/Test | Control2/Test/Control1
Started | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Visits 2, 3 and 4 - Period 1
Arm/Group | Test/Control1 | Control1/Test | Test/Control2 | Control2/Test | Test/Control1/Control2 | Test/Control2/Control1 | Control1/Control2/Test | Control1/Test/Control2 | Control2/Control1/Test | Control2/Test/Control1
Started | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Visits 2, 3 and 4 - Period 2
Arm/Group | Test/Control1 | Control1/Test | Test/Control2 | Control2/Test | Test/Control1/Control2 | Test/Control2/Control1 | Control1/Control2/Test | Control1/Test/Control2 | Control2/Control1/Test | Control2/Test/Control1
Started | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Visits 2, 3 and 4 - Period 3
Arm/Group | Test/Control1 | Control1/Test | Test/Control2 | Control2/Test | Test/Control1/Control2 | Test/Control2/Control1 | Control1/Control2/Test | Control1/Test/Control2 | Control2/Control1/Test | Control2/Test/Control1
Started | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9
  White | 13
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Nighttime Driving Score
Description: Overall driving performance score is a composite score calculated as the mean of the Z-scores of the following six driving measures: average sign recognition distance (in meters), percentage of correctly identified sign (~42 signs), percentage of hazard avoidance/detection (9 hazards), average pedestrian recognition distance (in meters), lane keeping (percentage of time inside the lane) and the inverse of driving lap time (in seconds).). Equal weighting was assigned to each measure. The individual Z scores were transformed (inverted) such that positive Z scores relate to better performance than the mean. Z scores follow a standard normal distribution (ranging from minus infinity to positive infinity). Overall Z score for night time driving was reported for each study lens.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol violation.
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- Test: Subjects that wore the Test lens during any of the three study periods at either visit 3 or visit 4.
- Control 1: Subjects that wore the Control 1 lens during any of the three study periods at either visit 3 or visit 4.
- Control 2: Subjects that wore the Control 2 lens during any of the three study periods at either visit 3 or visit 4.
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
Z-Score | -0.308 (0.4718) | -0.375 (0.4361) | -0.430 (0.4761)
Statistical Analysis 1: Comparison: Test vs Control 1; It was calculated that a total of 24 participants was required to show that the Test lens is non-inferior to the control 1 lens with 80% power. Sample size for this study was based on night driving only; Test type: Non-Inferiority — A non-inferiority margin of -0.25 was used. Non-inferioirty was concluded if the lower limit of the 95% CI was above 0.25; Linear Mixed Model; Kenward and Roger Method was used for denominator degrees of freedom; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [-0.045 to 0.183], Standard Error of Mean 0.0574 — Mean difference was calculated as Test - Control 1

2. Secondary Outcome: Binocular Visual Acuity
Description: Binocular visual acuity was assessed under Low luminance (~1 lux) high contrast (90%) conditions at a distance of 4 meters. The ETDRS logMAR chart were used, which is scored on a letter by letter basis (-0.02 log units per letter correctly identified). A number of different EDTRS charts was used to reduce potential learning effects. The average LogMAR acuity for each lens was reported.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
logMAR | 0.251 (0.0722) | 0.273 (0.0705) | 0.298 (0.0739)
Statistical Analysis 1: Comparison: Test vs Control 1; Test type: Non-Inferiority — A non-inferiority margin of 0.1 logMAR was used. Non-inferiority was concluded if the upper limit was below 0.1; Linear Mixed Model; Kenward and Roger Method was used for the degrees of freedom; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.043 to -0.012], Standard Error of Mean 0.0076 — Mean difference was calculated as Test - Control 1

3. Secondary Outcome: Binocular Contrast Threshold Without Glare
Description: Binocular contrast sensitivity was assessed under low luminance conditions. Five Landolt C targets in random orientation were presented for each of the four contrast levels 95%, 80%, 63% and 50%. Participants were asked to correctly identify the orientation of the Landolt C. The percentage of subjects that were able to correct identify the orientation of all 5 Landolt's C was reported for each lens type.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
Percentage of Participants
  95% Contrast | 100 | 100 | 100
  80% Contrast | 100 | 95.8 | 95.8
  63% Contrast | 91.7 | 91.7 | 87.5
  50% | 87.5 | 75.0 | 58.3
Statistical Analysis 1: Comparison: Test vs Control 1; Test type: Equivalence — Equivalence was concluded if 0 was contained in the 95% confidence interval; Generalized Estimating Equation; Odds Ratio (OR) = 3.162, 95% CI 2-sided [0.442 to 22.604] — Odds ratio was calculated as Test over Control 1

4. Secondary Outcome: Percentage of Road Signs Correctly Identified During Night Driving
Description: Participants were instructed to report the identity of a percentage of the standard road signs (typically about 42 signs dependent on the route travelled) containing about 65 items of information as they drove around the circuit. The percentage of correctly identified signs was reported for each study lens.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
Percentage of participants | 72.7 | 73.3 | 73.3
Statistical Analysis 1: Comparison: Test vs Control 1; Test type: Equivalence — Equivalence was concluded if 0 was contained in the 95% confidence interval; Generalized Linear Mixed Model; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.82 to 1.16] — Odds ratio was calculated as Test over Control1

5. Secondary Outcome: Average Distance to Correctly Identify Road Signs During Night Driving
Description: Measure Description The distance (measured in meters) to recognize a pre-determined road sign was recorded for each subject and lens type at either visit 3 or visit 4, using the in-vehicle measurement system while the participant was driving. The in-vehicle measurement system consisted of a subject pressing a button once the subject was able to recognize the road sign. The average distance in meters was reported for each lens type. Larger distance indicate that a subject was able to identify the pre-determined road sign sooner.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
Meters | 110.3 (23.45) | 101.5 (25.53) | 95.0 (22.83)
Statistical Analysis 1: Comparison: Test vs Control 1; Test type: Equivalence — Equivalence was concluded if 0 was contained in the 95% confidence interval; Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Mean Difference (Final Values) = 17.8, 95% CI 2-sided [7.1 to 28.5], Standard Error of Mean 5.29 — Mean difference was calculated as Test - Control 1

6. Secondary Outcome: Percentage of Hazards Avoided During Night Driving
Description: Participants were required to report and avoid hitting any of nine large, low contrast grey foam "hazards" (220 cm x 80 cm x 15 cm) positioned orthogonally in the driving lane along the roadway, the locations of which will be randomized between study lenses. The percentage of Hazards avoided for each study lens was reported.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
Percentage of Participants | 95.4 | 95.4 | 93.1
Statistical Analysis 1: Comparison: Test vs Control 1; Test type: Equivalence — Equivalence was concluded if 0 was contained in the 95% confidence interval; Generalized Linear Mixed Model; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.33 to 1.74] — Odds Ratio was calculated as Test over Control 1

7. Secondary Outcome: Average Pedestrian Recognition Distance
Description: The in-vehicle measurement system was utilized to determine the distance at which the participant (as a driver) first recognizes the presence of two pedestrians positioned at the side of the road. An experimenter acted as the pedestrian and "walked in-place" at the end of a 400 m straight section of roadway which starts and finishes at approximately the same elevation, but features a dip halfway along its length. The pedestrian was not surrounded by any visual clutter or lighting. To reduce expectancy effects, a series of four flashing LEDs and four retro-reflective bollards was positioned around the circuit to increase the instances of flashing lights and retro-reflective material being presented to the driver. The average distance to recognize a pedestrian for each lens type was reported.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 24 | 24 | 24
Meters | 208.3 (60.46) | 201.1 (62.92) | 195.5 (60.70)
Statistical Analysis 1: Comparison: Test vs Control 1; Test type: Equivalence — Equivalence was concluded if 0 was contained in the 95% confidence interval; Linear Mixed Model; Kenward and Roger Method was used for denominator Degrees of Freedom; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-11.4 to 20.7], Standard Error of Mean 7.93 — Mean difference was calculated as Test - Control 1

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 2 weeks per subject.
Groups:
- Control 1: Subjects that wore the Control 1 lens at any point in the study.
- Control 2: Subjects that wore the Control lens at any point in the study.
- Test: Subjects that wore the Test lens at any point in the study.
Arm/Group | Control 1 | Control 2 | Test
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03330275/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03330275/SAP_001.pdf